CLINICAL TRIAL: NCT03814551
Title: Young Adult Beverage and Health Study
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of California, Berkeley (Other)
Responsible Party: Sponsor
Other Study IDs: 1124060-2; 1K01DK113068-01A1 (NIH)
Record Dates: First submitted 2019-01-18; First posted 2019-01-24 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Comparison: Cohort of participants who regularly eat in cafeteria without health signage.
- Signage: Cohort of participants who regularly eat in cafeteria in which health signage is placed.
  Interventions: Behavioral: Signage

INTERVENTIONS:
Behavioral: Signage — Placement of signage discouraging consumption of beverages with added sugar
  Groups: Signage

SUMMARY:
This study examines the impact of health signage on beverage consumption in a cafeteria.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate student or staff member at specific university
* Age 18+
* On meal plan if a student
* Works in specific cafeterias if staff

Exclusion Criteria:

* Age <18 years
* Adults unable to consent or complete the written or online survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At specific university: Undergraduate college students on meal plan and university staff
Sampling Method: Non-Probability Sample
Enrollment: 911 (Actual)
Dates: Start 2018-11-24 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Change in self-reported sugar-sweetened beverage consumption | 5 months
  Beverage frequency questionnaire assessing whether various beverages were consumed "4 or more times per day," "3 times per day," "2 times per day," "1 time per day," "4-6 times per week," "2-3 times per week," "one time per week or less," or "never" in the last/current semester.

SECONDARY OUTCOMES:
Change in cafeteria sugar-sweetened beverage usage | 5 months
  Based on inventory and syrup/beverage purchase data and customer counts.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Falbe, ScD, MPH, Principal Investigator — UC Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No